CLINICAL TRIAL: NCT06609772
Title: The Effect of Individualised Pain Education on Chronic Postoperative Pain Development and Quality of Life in Living Liver Donors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazlican Bagci (Other)
Responsible Party: Sponsor-Investigator, Nazlican Bagci, PhD student, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024/6148
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Quality of Life; Living-donor Liver Transplantation; Chronic Post Operative Pain; Pain Management
Keywords: Living Liver Donors; Chronic Postoperative Pain; Individualised Pain Education; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: Power analysis was performed to calculate the sample size of this study. According to the calculation made using the G*power 3.1 program; the sample size was determined as 110 (55 experimental, 55 control) with an effect size of 0.22, a margin of error of 0.05, a confidence level of 0.95, and a universe representation power of 0.95. Considering the possible losses that may occur for any reason, it was planned to include 120 individuals (60 experimental, 60 control) who are living liver donors in the study. In this study, the randomization method will be used in assigning the participants to the control and experimental groups. Thus, it was aimed to protect the randomization in case of data loss. Computer-assisted randomization will be used for randomization.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): After obtaining the necessary legal and ethical permissions for data collection, the research will commence. During this stage of the study, participants who agree to take part in the research will be asked to fill out the informed consent form. To obtain the pre-test data for the research, all forms will be filled out. The patients will be called by the researcher on the 15th, 45th and 75th days to perform interim measurements (Interim measurement-1, Interim measurement-2, Interim measurement-3). On the 90th and 120th days, the patients will be called again by the researcher and the final tests will be applied.
- Individualized pain education group (Experimental): During this stage of the study, participants who agree to take part in the research will be asked to fill out the informed consent form. The individualized pain education program is planned to be applied to all patients on the 6th postoperative day. To obtain the pre-test data for the research, all forms will be filled out. Individual education will be given to the patients in the experimental group in their own rooms and all questions asked by the patient will be answered after the education. The education booklet will be given to the patients after the individual education program. The patients in the experimental group will be informed that they will be called via video call for the 30th and 60th day reminder education. The patients will be called by the researcher on the 15th, 45th and 75th days to perform interim measurements. On the 90th and 120th days, the patients will be called again by the researcher and the final tests will be applied.
  Interventions: Other: Individualised Pain Education

INTERVENTIONS:
Other: Individualised Pain Education — Individualised Pain Education
  Arms: Individualized pain education group

SUMMARY:
Chronic postoperative pain is defined as pain that is a continuation of acute pain or develops after a pain-free period, is localised to the surgical site, affects quality of life, and persists for at least 3 months after surgery when other pain factors are excluded. Chronic postoperative pain, as a major complication of surgery, increases the use of analgesics, restricts activities of daily living, reduces quality of life and creates a serious economic burden. Prolonged pain in the preoperative period and poorly treated postoperative acute pain may trigger the development of chronic pain. Chronic postoperative pain is an important and current problem in living liver transplant donors as in many patient groups.

Chronic pain due to severe postoperative acute pain is reported as an expected outcome after open surgical resection in living liver transplant donors. The reason for this is thought to be inadequate perioperative pain management. Inadequate perioperative pain management may lead to sub-optimal pain management, delayed recovery, unexpected readmissions, decreased patient satisfaction, prolonged duration of opioid analgesia with potential for narcotic abuse, and clinical, psychological and socioeconomic consequences that may possibly lead to chronic postoperative pain. Chronic postoperative pain is a common but overlooked complication of surgery that can cause functional limitation, psychological distress and poor quality of life in patients and its management is very important for nurses. An important aim of nursing care is to help liver living donors regain their health and quality of life. Providing management of acute postoperative pain, preventing the development of chronic postoperative pain and improving quality of life in patients undergoing surgical procedures are important issues for nurses. At the same time, chronic postoperative pain management, as a very current issue, requires nurses to plan and implement more effective interventions. With appropriate pain interventions in the preoperative and early postoperative period, the patient should be educated and counselled about self-management strategies, return to normal functionality and the possibility of developing chronic pain after surgery. Adequate perioperative education about the surgery and expected outcomes may alleviate stress, reduce the severity of acute pain and help prevent chronic postoperative pain.

It is thought that individualised pain education will be effective on chronic postoperative pain development and quality of life of patients. When the literature was reviewed, no study on individualised pain education for liver living donors was found. At the same time, no study was found in the literature in which chronic postoperative pain and quality of life were examined together in liver living donors. The fact that the subject will be investigated for the first time adds originality to the study.

With this study, the effect of individualised pain education on prevention or reduction of chronic postoperative pain and improvement of quality of life will be determined. Thus, the data obtained can be evaluated holistically and can form the basis for new and large-scale studies in the related field. At the same time, in this prospective study, the rates and characteristics of chronic postoperative pain development in liver living donors at the 3rd month after transplantation will be evaluated. Thus, this study will contribute to the limited literature on this subject.

Research Hypotheses:

H0a: Individualized pain education applied to living liver donors is not effective on the development of chronic postoperative pain.

H1a: Individualized pain education applied to living liver donors is effective on the development of chronic postoperative pain.

H0b: Individualized pain education applied to living liver donors is not effective on the quality of life of patients.

H1b: Individualized pain education applied to living liver donors is effective on the quality of life of patients.

DETAILED DESCRIPTION:
Chronic postoperative pain is defined as pain that is a continuation of acute pain or develops after a pain-free period, is localised to the surgical site, affects quality of life, and persists for at least 3 months after surgery when other pain factors are excluded. As a common condition, it affects approximately 5% to 85% of all surgical patients. Chronic postoperative pain, as a major complication of surgery, increases the use of analgesics, restricts activities of daily living, reduces quality of life and creates a serious economic burden. It also causes negative consequences such as anxiety, depression, sleep disorders and opioid use disorders. Prolonged pain in the preoperative period and poorly treated postoperative acute pain may trigger the development of chronic pain. It has also been reported that factors such as young age, female gender, high body mass index, smoking, fear, anxiety, and duration of surgery may be associated with chronic postoperative pain. Chronic postoperative pain is an important and current problem in living liver transplant donors as in many patient groups. Although limited data are available, some studies report that donors experience chronic pain beyond the expected normal recovery period.

Chronic pain due to severe postoperative acute pain is reported as an expected outcome after open surgical resection in living liver transplant donors. The reason for this is thought to be inadequate perioperative pain management. Inadequate perioperative pain management may lead to sub-optimal pain management, delayed recovery, unexpected readmissions, decreased patient satisfaction, prolonged duration of opioid analgesia with potential for narcotic abuse, and clinical, psychological and socioeconomic consequences that may possibly lead to chronic postoperative pain. Chronic postoperative pain is a common but overlooked complication of surgery that can cause functional limitation, psychological distress and poor quality of life in patients and its management is very important for nurses. An important aim of nursing care is to help liver living donors regain their health and quality of life. Providing management of acute postoperative pain, preventing the development of chronic postoperative pain and improving quality of life in patients undergoing surgical procedures are important issues for nurses. At the same time, chronic postoperative pain management, as a very current issue, requires nurses to plan and implement more effective interventions. With appropriate pain interventions in the preoperative and early postoperative period, the patient should be educated and counselled about self-management strategies, return to normal functionality and the possibility of developing chronic pain after surgery. Adequate perioperative education about the surgery and expected outcomes may alleviate stress, reduce the severity of acute pain and help prevent chronic postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* No condition that prevents communication
* Having the ability to read and write
* No major complications in the early postoperative period
* No previous abdominal surgery
* No additional disease that may cause chronic pain

Exclusion Criteria:

* Having any condition that prevents communication
* Lack of reading and writing skills
* Having a major complication in the early postoperative period
* Having had abdominal surgery before
* Having an additional disease that may cause chronic pain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Chronic Postoperative Pain Development | 120 days
  Whether Chronic Postoperative Pain develops or not will be evaluated using the numeric rating scale (NRS). In NRS, the patient is asked to give a numerical score for their pain between 0 and 10 or 0 and 100. On the scale, 0 indicates no pain, 1-3 indicates mild pain, 4-6 indicates moderate pain, and 7-10 indicates severe pain. NRS is an easy and understandable method.
Chronic Postoperative Pain Development | 120 days
  In the presence of Chronic Postoperative Pain, the pain will be assessed using the McGill-Melzack Pain Questionnaire (MASF). With the scale; the location of the pain in the first part, the characteristics of the pain in the second part, the variables that reduce and increase the pain in the third part and the severity of the pain in the fourth part. The total score is calculated in the scale (0-112).
Quality of Life | 120 days
  It Quality of Life will be assessed using the EuroQol 5-Dimensional 3-Level (EQ-5D-3L) General Quality of Life Scale.
  The EQ-5D consists of a thermometer-like visual analog scale (EQ-VAS) anchored by 0 (worst health) and 100 (best health) to assess health status at the time of assessment and a 5-item descriptive system with five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has three levels of responses reflecting no, moderate, and extreme problems. The response pattern in these 5 items can be converted into a single index score, anchored between zero (for death) and 1 (perfect health).

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University Liver Transplant Institute, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This research is a doctoral thesis study. The research is expected to be completed.